CLINICAL TRIAL: NCT02370498
Title: A Phase III, Randomized, Open-label Clinical Trial of Pembrolizumab (MK-3475) Versus Paclitaxel in Subjects With Advanced Gastric or Gastroesophageal Junction Adenocarcinoma Who Progressed After First-Line Therapy With Platinum and Fluoropyrimidine
Brief Title: A Study of Pembrolizumab (MK-3475) Versus Paclitaxel for Participants With Advanced Gastric/Gastroesophageal Junction Adenocarcinoma That Progressed After Therapy With Platinum and Fluoropyrimidine (MK-3475-061/KEYNOTE-061)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-061; 152988 (Registry Identifier: JAPIC); MK-3475-061 (Other: Merck Protocol Number); 2014-005241-45 (EudraCT Number)
Record Dates: First submitted 2015-02-23; First posted 2015-02-25 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-05

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
Keywords: Gastric cancer; Gastroesophageal junction cancer; PD1; PD-1; PDL1; PD-L1
MeSH Terms: conditions — Stomach Neoplasms | interventions — pembrolizumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab (Experimental): Participants receive 200 mg intravenous (IV) pembrolizumab on Day 1 of each 21-day cycle, for up to 35 administrations (approximately 2 years).
  Interventions: Biological: pembrolizumab
- Paclitaxel (Active Comparator): Participants receive 80 mg/m^2 IV paclitaxel on Days 1, 8, and 15 of each 28-day cycle, until disease progression or unacceptable toxicity.
  Interventions: Drug: paclitaxel

INTERVENTIONS:
Biological: pembrolizumab — 200 mg administered as IV infusion on Day 1 of each 21-day cycle.
  Other Names: MK-3475
  Arms: Pembrolizumab
Drug: paclitaxel — 80 mg/m^2 administered as IV infusion on Days 1, 8, and 15 of each 28-day cycle.
  Other Names: TAXOL®
  Arms: Paclitaxel

SUMMARY:
This is a study for participants with advanced gastric or gastroesophageal junction adenocarcinoma who have had tumor progression after first-line treatment with platinum and fluoropyrimidine doublet therapy. The primary study hypotheses are that pembrolizumab (MK-3475) prolongs progression free survival (PFS) and overall survival (OS) for participants with tumors that show positive programmed cell death ligand 1 (PD-L1) expression.

As of 20-March-2016, enrollment will be limited to PD-L1 positive participants.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically-confirmed diagnosis of gastric or gastroesophageal junction adenocarcinoma
* Confirmed metastatic or locally advanced, unresectable disease (by computed tomography [CT] scan or clinical evidence)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Progression on or after prior first-line therapy containing any platinum/fluoropyrimidine doublet
* Willing to provide tumor tissue for PD-L1 biomarker analysis (new or archived specimens with agreement of Sponsor). As of 20 March 2016, participants must be PD-L1 positive to be enrolled.
* Human epidermal growth factor receptor 2 (HER-2/neu) status known and participants with HER2/neu positive tumors show documentation of disease progression on treatment containing trastuzumab
* Female participants of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of pembrolizumab or through 180 days after the last dose of paclitaxel.
* Male participants should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of pembrolizumab or through 180 days after the last dose of paclitaxel.
* Adequate organ function

Exclusion Criteria:

* Currently participating and receiving study therapy, or participated in a study of an investigational agent and received study therapy or used an investigation device within 4 weeks of the first dose of medication
* Squamous cell or undifferentiated gastric cancer
* Active autoimmune disease that has required systemic treatment in past 2 years (replacement therapy is not considered a form of systemic treatment
* Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study medication
* Prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or not recovered from AEs due to agents administered more than 4 weeks earlier
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or not recovered from adverse events due to a previously administered agent or surgery
* Known additional malignancy that is progressing or requires active treatment (with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy)
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* History of (noninfectious) pneumonitis that required steroids or current pneumonitis
* Active infection requiring systemic therapy
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of pembrolizumab or through 180 days after the last dose of paclitaxel.
* Prior immunotherapy including anti-PD-1, anti-PD-L1, or anti-PD-L2 agent, or previously participated in Merck pembrolizumab (MK-3475) clinical trial
* Known history of human immunodeficiency virus (HIV)
* Known active Hepatitis B or Hepatitis C
* Live vaccine within 30 days of planned start of study therapy
* Known allergy or hypersensitivity to paclitaxel or any components used in the paclitaxel preparation or other contraindication for taxane therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 592 (Actual)
Dates: Start 2015-05-11 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2021-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Janjigian YY, Cecchini M, Shitara K, Enzinger PC, Wainberg ZA, Chau I, Satoh T, Lee J, Nebozhyn M, Loboda A, Kobie J, Vajdi A, Shih CS, Cristescu R, Cao ZA. Genomic Landscape of Late-Stage Gastric Cancer: Analysis From KEYNOTE-059, KEYNOTE-061, and KEYNOTE-062 Studies. JCO Precis Oncol. 2025 Mar;9:e2400456. doi: 10.1200/PO-24-00456. Epub 2025 Mar 21. PMID 40117530
- [Derived] Shitara K, Di Bartolomeo M, Mandala M, Ryu MH, Caglevic C, Olesinski T, Chung HC, Muro K, Goekkurt E, McDermott RS, Mansoor W, Wainberg ZA, Shih CS, Kobie J, Nebozhyn M, Cristescu R, Cao ZA, Loboda A, Ozguroglu M. Association between gene expression signatures and clinical outcomes of pembrolizumab versus paclitaxel in advanced gastric cancer: exploratory analysis from the randomized, controlled, phase III KEYNOTE-061 trial. J Immunother Cancer. 2023 Jun;11(6):e006920. doi: 10.1136/jitc-2023-006920. PMID 37399357
- [Derived] Muro K, Shitara K, Yamaguchi K, Yoshikawa T, Satake H, Hara H, Sugimoto N, Machida N, Goto M, Kawakami H, Amagai K, Omuro Y, Esaki T, Hironaka S, Nishina T, Komatsu Y, Matsubara H, Shiratori S, Han S, Satoh T, Ohtsu A. Efficacy of Pembrolizumab Monotherapy in Japanese Patients with Advanced Gastric or Gastroesophageal Junction Cancer. J Gastrointest Cancer. 2023 Sep;54(3):951-961. doi: 10.1007/s12029-023-00920-9. Epub 2023 Apr 10. PMID 37037952
- [Derived] Cristescu R, Aurora-Garg D, Albright A, Xu L, Liu XQ, Loboda A, Lang L, Jin F, Rubin EH, Snyder A, Lunceford J. Tumor mutational burden predicts the efficacy of pembrolizumab monotherapy: a pan-tumor retrospective analysis of participants with advanced solid tumors. J Immunother Cancer. 2022 Jan;10(1):e003091. doi: 10.1136/jitc-2021-003091. PMID 35101941
- [Derived] Fuchs CS, Ozguroglu M, Bang YJ, Di Bartolomeo M, Mandala M, Ryu MH, Fornaro L, Olesinski T, Caglevic C, Chung HC, Muro K, Van Cutsem E, Elme A, Thuss-Patience P, Chau I, Ohtsu A, Bhagia P, Wang A, Shih CS, Shitara K. Pembrolizumab versus paclitaxel for previously treated PD-L1-positive advanced gastric or gastroesophageal junction cancer: 2-year update of the randomized phase 3 KEYNOTE-061 trial. Gastric Cancer. 2022 Jan;25(1):197-206. doi: 10.1007/s10120-021-01227-z. Epub 2021 Sep 1. PMID 34468869
- [Derived] Van Cutsem E, Amonkar M, Fuchs CS, Alsina M, Ozguroglu M, Bang YJ, Chung HC, Muro K, Goekkurt E, Benson AB 3rd, Sun W, Wainberg ZA, Norquist JM, Chen X, Shih CS, Shitara K. Health-related quality of life in advanced gastric/gastroesophageal junction cancer with second-line pembrolizumab in KEYNOTE-061. Gastric Cancer. 2021 Nov;24(6):1330-1340. doi: 10.1007/s10120-021-01200-w. Epub 2021 Aug 7. PMID 34363528
- [Derived] Chao J, Fuchs CS, Shitara K, Tabernero J, Muro K, Van Cutsem E, Bang YJ, De Vita F, Landers G, Yen CJ, Chau I, Elme A, Lee J, Ozguroglu M, Catenacci D, Yoon HH, Chen E, Adelberg D, Shih CS, Shah S, Bhagia P, Wainberg ZA. Assessment of Pembrolizumab Therapy for the Treatment of Microsatellite Instability-High Gastric or Gastroesophageal Junction Cancer Among Patients in the KEYNOTE-059, KEYNOTE-061, and KEYNOTE-062 Clinical Trials. JAMA Oncol. 2021 Jun 1;7(6):895-902. doi: 10.1001/jamaoncol.2021.0275. PMID 33792646
- [Derived] Shitara K, Ozguroglu M, Bang YJ, Di Bartolomeo M, Mandala M, Ryu MH, Fornaro L, Olesinski T, Caglevic C, Chung HC, Muro K, Goekkurt E, Mansoor W, McDermott RS, Shacham-Shmueli E, Chen X, Mayo C, Kang SP, Ohtsu A, Fuchs CS; KEYNOTE-061 investigators. Pembrolizumab versus paclitaxel for previously treated, advanced gastric or gastro-oesophageal junction cancer (KEYNOTE-061): a randomised, open-label, controlled, phase 3 trial. Lancet. 2018 Jul 14;392(10142):123-133. doi: 10.1016/S0140-6736(18)31257-1. Epub 2018 Jun 4. PMID 29880231
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After 20 March 2016, enrollment was limited to programmed cell death ligand 1 (PD-L1) positive participants.
Pre-assignment Details: Of 592 participants that were randomized to trial, 570 received treatment. At the time of the primary analysis data cut-off, 89 participants are ongoing in the study.
Groups:
- Paclitaxel: Participants receive paclitaxel 80 mg/m^2 IV, on Days 1, 8, and 15 of each 28-day cycle until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Pembrolizumab | Paclitaxel
Started | 296 | 296
Treated | 294 | 276
PD-L1 Positive Participants | 196 | 199
Completed | 0 | 0
Not Completed | 296 | 296
Not completed — Adverse Event | 10 | 8
Not completed — Death | 263 | 265
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 7 | 12
Not completed — Sponsor's decision | 15 | 9

BASELINE CHARACTERISTICS:
Groups:
- Pembrolizumab: Participants receive 200 mg IV pembrolizumab on Day 1 of each 21-day cycle, for up to 35 administrations (approximately 2 years).
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab | Paclitaxel | Total
Number analyzed (Participants) | 296 | 296 | 592
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.7 (12.0) | 59.6 (11.7) | 60.2 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 88 | 182
  Male | 202 | 208 | 410
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 24 | 51
  Not Hispanic or Latino | 269 | 272 | 541
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 7
  Asian | 93 | 91 | 184
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 193 | 198 | 391
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  Europe/Israel/North America/Australia | 190 | 187 | 377
  Asia | 88 | 89 | 177
  Rest of World | 18 | 20 | 38
PD-L1 Status [Count of Participants; unit: Participants]
  Positive | 196 | 199 | 395
  Negative | 99 | 96 | 195
  Unknown | 1 | 1 | 2
Time To Progression (TTP) on first-line therapy [Count of Participants; unit: Participants]
  <6 months | 186 | 182 | 368
  ≥6 months | 110 | 114 | 224

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) According to Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1) Based on Blinded Independent Central Review (BICR) in Programmed Death-Ligand 1 (PD-L1) Positive Participants
Description: PFS was defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on BICR, or death due to any cause, whichever occurs first. According to RECIST 1.1, progressive disease (PD) was defined as a 20% relative increase in the sum of diameters (SOD) of target lesions, taking as reference the nadir SOD and an absolute increase of >5 mm in the SOD, or the appearance of new lesions. PFS was analyzed using the Kaplan-Meier method and median PFS (95% confidence interval [CI]) in months was reported for PD-L1 positive participants by treatment group.
Time Frame: Up to 30 months (through database cut-off date of 26 Oct 2017)
Population: All randomized PD-L1 positive participants. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab | Paclitaxel
Number analyzed (Participants) | 196 | 199
months | 1.5 [1.4 to 2.0] | 4.1 [3.1 to 4.2]
Statistical Analysis 1: Comparison: Pembrolizumab vs Paclitaxel; Treatment difference in PFS was assessed by the Stratified Log-rank test, and a stratified Cox proportional hazard model with Efron's method of tie handling was used to assess the magnitude of the treatment difference (Hazard Ratio [HR]) between the treatment arms; Test type: Other; p = 0.98358, Regression, Cox — One-sided p-value based on log-rank test stratified by geographic region (Europe/Israel/North America/Australia vs. Asia vs. Rest of World) and TTP on first-line therapy (< 6 months vs. >= 6 months); P-value rounded to 5 decimal places; Hazard Ratio (HR) = 1.27, 95% CI 2-sided [1.03 to 1.57]

2. Primary Outcome: Overall Survival (OS) in PD-L1 Positive Participants
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. OS was analyzed using the Kaplan-Meier method and median OS (95% CI) in months was reported for PD-L1 positive participants by treatment group.
Time Frame: Up to 30 months (through database cut-off date of 26 Oct 2017)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab | Paclitaxel
Number analyzed (Participants) | 196 | 199
months | 9.1 [6.2 to 10.7] | 8.3 [7.6 to 9.0]
Statistical Analysis 1: Comparison: Pembrolizumab vs Paclitaxel; Treatment difference in OS was assessed by the Stratified Log-rank test, and a stratified Cox proportional hazard model with Efron's method of tie handling was used to assess the magnitude of the treatment difference (HR) between the treatment arms; Test type: Other; p = 0.04205, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; P-value rounded to 5 decimal places; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.66 to 1.03]

3. Secondary Outcome: PFS According to RECIST 1.1 Based on BICR in All Participants
Description: PFS was defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on BICR, or death due to any cause, whichever occurs first. According to RECIST 1.1, PD was defined as a 20% relative increase in the SOD of target lesions, taking as reference the nadir SOD and an absolute increase of >5 mm in the SOD, or the appearance of new lesions. PFS was analyzed using the Kaplan-Meier method and median PFS (95% CI) in months was reported for all participants by treatment group.
Time Frame: Up to 30 months (through database cut-off date of 26 Oct 2017)
Population: All randomized participants. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab | Paclitaxel
Number analyzed (Participants) | 296 | 296
months | 1.5 [1.4 to 1.6] | 4.1 [3.2 to 4.2]
Statistical Analysis 1: Comparison: Pembrolizumab vs Paclitaxel; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.99999, Regression, Cox — One-sided p-value based on log-rank test stratified by geographic region (Europe/Israel/North America/Australia vs. Asia vs. Rest of World), TTP on first-line therapy (< 6 months vs. >= 6 months), and PD-L1 status (positive vs. negative); P-value rounded to 5 decimal places; Hazard Ratio (HR) = 1.49, 95% CI 2-sided [1.25 to 1.77]

4. Secondary Outcome: OS in All Participants
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. OS was analyzed using the Kaplan-Meier method and median OS (95% CI) in months was reported for all participants by treatment group.
Time Frame: Up to 30 months (through database cut-off date of 26 Oct 2017)
Population: All randomized participants. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab | Paclitaxel
Number analyzed (Participants) | 296 | 296
months | 6.7 [5.4 to 8.9] | 8.3 [7.7 to 8.8]
Statistical Analysis 1: Comparison: Pembrolizumab vs Paclitaxel; Treatment difference in OS was assessed by the Stratified Log-rank test, and a stratified Cox proportional hazard model with Efron's method of tie handling was used to assess the magnitude of the treatment difference (Hazard Ratio [HR]) between the treatment arms; Test type: Other; p = 0.24463, Regression, Cox — One-sided p-value based on log-rank test stratified by geographic region (Europe/Israel/North America/Australia vs. Asia vs. Rest of World), TTP on first-line therapy (<6 months vs. ≥6 months), and PD-L1 status (positive vs. negative); P-value rounded to 5 decimal places; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.79 to 1.12]

5. Secondary Outcome: PFS According to RECIST 1.1 Based on Investigator Assessment in PD-L1 Positive Participants
Description: PFS was defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on investigator assessment, or death due to any cause, whichever occurs first. According to RECIST 1.1, PD was defined as a 20% relative increase in the SOD of target lesions, taking as reference the nadir SOD and an absolute increase of >5 mm in the SOD, or the appearance of new lesions. PFS was analyzed using the Kaplan-Meier method and median PFS (95% CI) in months was reported for PD-L1 positive participants by treatment group.
Time Frame: Up to 30 months (through database cut-off date of 26 Oct 2017)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab | Paclitaxel
Number analyzed (Participants) | 196 | 199
months | 1.6 [1.5 to 2.7] | 3.1 [2.8 to 4.0]
Statistical Analysis 1: Comparison: Pembrolizumab vs Paclitaxel; Treatment difference in PFS was assessed by the Stratified Log-rank test, and a stratified Cox proportional hazard model with Efron's method of tie handling was used to assess the magnitude of the treatment difference (HR) between the treatment arms; Test type: Other; p = 0.41331, Regression, Cox — One-sided p-value based on log-rank test stratified by geographic region (Europe/Israel/North America/Australia vs. Asia vs. Rest of World) and TTP on first-line therapy (<6 months vs. ≥6 months); P-value rounded to 5 decimal places; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.79 to 1.21]

6. Secondary Outcome: PFS According to RECIST 1.1 Based on Investigator Assessment in All Participants
Description: PFS was defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on investigator assessment, or death due to any cause, whichever occurs first. According to RECIST 1.1, PD was defined as a 20% relative increase in the SOD of target lesions, taking as reference the nadir SOD and an absolute increase of >5 mm in the SOD, or the appearance of new lesions. PFS was analyzed using the Kaplan-Meier method and median PFS (95% CI) in months was reported for all participants by treatment group.
Time Frame: Up to 30 months (through database cut-off date of 26 Oct 2017)
Population: All randomized participants. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab | Paclitaxel
Number analyzed (Participants) | 296 | 296
months | 1.6 [1.5 to 1.9] | 3.2 [2.9 to 4.0]
Statistical Analysis 1: Comparison: Pembrolizumab vs Paclitaxel; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.97481, Regression, Cox — [p-value comment as in outcome 4, analysis 1]; P-value rounded to 5 decimal places; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [1.00 to 1.42]

7. Secondary Outcome: PFS According to Immune-Related Response Evaluation Criteria in Solid Tumors (irRECIST) Based on BICR in PD-L1 Positive Participants
Description: PFS defined as time from randomization to first documented PD per irRECIST based on BICR, or death due to any cause, whichever occurs first. Following initial PD by RECIST 1.1 (20% relative increase in SOD of target lesions), participants were assessed according to irRECIST: tumor assessment was repeated ≥4 weeks later to confirm PD with the option of continuing treatment until this scan was obtained for clinically stable participants. If PD confirmed, participant was discontinued from treatment unless investigator determined benefit. If repeat scan indicated stable disease (SD; neither sufficient shrinkage or increase of target lesion), partial response (PR; ≥30% decrease in the SOD of target lesions), or complete response (CR; disappearance of all non-nodal target lesions), participant could continue treatment at investigator's discretion. PFS analyzed using Kaplan-Meier method and median PFS (95% CI) in months was reported for PD-L1 positive participants by treatment group.
Time Frame: Up to 30 months (through database cut-off date of 26 Oct 2017)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab | Paclitaxel
Number analyzed (Participants) | 196 | 199
months | 1.9 [1.4 to 3.0] | 4.2 [3.5 to 4.4]
Statistical Analysis 1: Comparison: Pembrolizumab vs Paclitaxel; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.80696, Regression, Cox — [p-value comment as in outcome 5, analysis 1]; P-value rounded to 5 decimal places; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.89 to 1.38]

8. Secondary Outcome: PFS According to irRECIST Based on BICR in All Participants
Description: PFS defined as time from randomization to first documented PD per irRECIST based on BICR, or death due to any cause, whichever occurs first. Following initial PD by RECIST 1.1 (20% relative increase in SOD of target lesions), participants were assessed according to irRECIST: tumor assessment was repeated ≥4 weeks later to confirm PD with the option of continuing treatment until this scan was obtained for clinically stable participants. If PD confirmed, participant was discontinued from treatment unless investigator determined benefit. If repeat scan indicated SD (neither sufficient shrinkage or increase of target lesion), PR (≥30% decrease in the SOD of target lesions), or CR (disappearance of all non-nodal target lesions), participant could continue treatment at investigator's discretion. PFS analyzed using Kaplan-Meier method and median PFS (95% CI) in months was reported for all participants by treatment group.
Time Frame: Up to 30 months (through database cut-off date of 26 Oct 2017)
Population: All randomized participants. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab | Paclitaxel
Number analyzed (Participants) | 296 | 296
months | 1.6 [1.5 to 2.5] | 4.2 [4.0 to 4.4]
Statistical Analysis 1: Comparison: Pembrolizumab vs Paclitaxel; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.99932, Regression, Cox — [p-value comment as in outcome 3, analysis 1]; P-value rounded to 5 decimal places; Hazard Ratio (HR) = 1.34, 95% CI 2-sided [1.12 to 1.60]

9. Secondary Outcome: Time to Tumor Progression (TTP) According to RECIST 1.1 Based on BICR in PD-L1 Positive Participants
Description: TTP was defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on BICR. Using RECIST 1.1, progressive disease was defined as a 20% relative increase in the SOD of target lesions, taking as reference the nadir SOD and an absolute increase of >5 mm in the SOD, or the appearance of new lesions. If there was no documented disease progression, TTP was censored at last tumor assessment date. TTP was analyzed using the Kaplan-Meier method and median TTP (95% CI) in months was reported for PD-L1 positive participants by treatment group.
Time Frame: Up to 30 months (through database cut-off date of 26 Oct 2017)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab | Paclitaxel
Number analyzed (Participants) | 196 | 199
months | 1.6 [1.4 to 2.7] | 4.0 [3.1 to 4.2]
Statistical Analysis 1: Comparison: Pembrolizumab vs Paclitaxel; Treatment difference in TTP was assessed by the Stratified Log-rank test, and a stratified Cox proportional hazard model with Efron's method of tie handling was used to assess the magnitude of the treatment difference (HR) between the treatment arms; Test type: Other; p = 0.99661, Regression, Cox — [p-value comment as in outcome 5, analysis 1]; P-value rounded to 5 decimal places; Hazard Ratio (HR) = 1.45, 95% CI 2-sided [1.11 to 1.89]

10. Secondary Outcome: TTP According to RECIST 1.1 Based on BICR in All Participants
Description: TTP was defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on BICR. Using RECIST 1.1, progressive disease was defined as a 20% relative increase in the SOD of target lesions, taking as reference the nadir SOD and an absolute increase of >5 mm in the SOD, or the appearance of new lesions. If there was no documented disease progression, TTP was censored at last tumor assessment date. TTP was analyzed using the Kaplan-Meier method and median TTP (95% CI) in months was reported for all participants by treatment group.
Time Frame: Up to 30 months (through database cut-off date of 26 Oct 2017)
Population: All randomized participants. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab | Paclitaxel
Number analyzed (Participants) | 296 | 296
months | 1.5 [1.4 to 1.8] | 4.1 [3.2 to 4.2]
Statistical Analysis 1: Comparison: Pembrolizumab vs Paclitaxel; [analysis description as in outcome 9, analysis 1]; Test type: Other; p = 1.00000, Regression, Cox — [p-value comment as in outcome 3, analysis 1]; P-value rounded to 5 decimal places; Hazard Ratio (HR) = 1.77, 95% CI 2-sided [1.42 to 2.20]

11. Secondary Outcome: TTP According to RECIST 1.1 Based on Investigator Assessment in PD-L1 Positive Participants
Description: TTP was defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on investigator assessment. Using RECIST 1.1, progressive disease was defined as a 20% relative increase in the SOD of target lesions, taking as reference the nadir SOD and an absolute increase of >5 mm in the SOD, or the appearance of new lesions. If there was no documented disease progression, TTP was censored at last tumor assessment date. TTP was analyzed using the Kaplan-Meier method and median TTP (95% CI) in months was reported for PD-L1 positive participants by treatment group.
Time Frame: Up to 30 months (through database cut-off date of 26 Oct 2017)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab | Paclitaxel
Number analyzed (Participants) | 196 | 199
months | 2.1 [1.5 to 3.0] | 3.3 [2.9 to 4.1]
Statistical Analysis 1: Comparison: Pembrolizumab vs Paclitaxel; [analysis description as in outcome 9, analysis 1]; Test type: Other; p = 0.39280, Regression, Cox — [p-value comment as in outcome 5, analysis 1]; P-value rounded to 5 decimal places; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.77 to 1.23]

12. Secondary Outcome: TTP According to RECIST 1.1 Based on Investigator Assessment in All Participants
Description: TTP was defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on investigator assessment. Using RECIST 1.1, progressive disease was defined as a 20% relative increase in the SOD of target lesions, taking as reference the nadir SOD and an absolute increase of >5 mm in the SOD, or the appearance of new lesions. If there was no documented disease progression, TTP was censored at last tumor assessment date. TTP was analyzed using the Kaplan-Meier method and median TTP (95% CI) in months was reported for all participants by treatment group.
Time Frame: Up to 30 months (through database cut-off date of 26 Oct 2017)
Population: All randomized participants. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab | Paclitaxel
Number analyzed (Participants) | 296 | 296
months | 1.6 [1.5 to 2.7] | 3.8 [3.0 to 4.1]
Statistical Analysis 1: Comparison: Pembrolizumab vs Paclitaxel; [analysis description as in outcome 9, analysis 1]; Test type: Other; p = 0.97033, Regression, Cox — [p-value comment as in outcome 3, analysis 1]; P-value rounded to 5 decimal places; Hazard Ratio (HR) = 1.21, 95% CI 2-sided [1.00 to 1.47]

13. Secondary Outcome: Objective Response Rate (ORR) According to RECIST 1.1 Based on BICR in PD-L1 Positive Participants
Description: ORR was defined as the percentage of the participants in the analysis population who had a confirmed CR (disappearance of all non-nodal target lesions and any pathological lymph nodes must have become normal) or PR (at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD) according to RECIST 1.1 and based on BICR. ORR was analyzed using the stratified Miettinen and Nurminen method, and reported with 95% CI for PD-L1 positive participants by treatment group.
Time Frame: Up to 30 months (through database cut-off date of 26 Oct 2017)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab | Paclitaxel
Number analyzed (Participants) | 196 | 199
Percentage of participants | 15.8 [11.0 to 21.7] | 13.6 [9.1 to 19.1]
Statistical Analysis 1: Comparison: Pembrolizumab vs Paclitaxel; Stratified Miettinen and Nurminen's (MN) method was used for comparison of the ORR between the treatment arms. A 95% CI for the difference in response rates between the pembrolizumab arm and paclitaxel arm was provided; Test type: Other; p = 0.28967, Miettinen and Nurminen method — Stratification factors for MN method included geographic region (Europe/Israel/North America/Australia vs. Asia vs. Rest of World) and TTP on first-line therapy (<6 months vs. ≥6 months) weighting by sample size; P-value rounded to 5 decimal places; Difference in Percentage = 2.0, 95% CI 2-sided [-5.0 to 9.1]

14. Secondary Outcome: ORR According to RECIST 1.1 Based on BICR in All Participants
Description: ORR was defined as the percentage of the participants in the analysis population who had a confirmed CR (disappearance of all non-nodal target lesions and any pathological lymph nodes must have become normal) or PR (at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD) according to RECIST 1.1 and based on BICR. ORR was analyzed using the stratified Miettinen and Nurminen method, and reported with 95% CI for all participants by treatment group.
Time Frame: Up to 30 months (through database cut-off date of 26 Oct 2017)
Population: All randomized participants. Participants were included in the treatment group to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab | Paclitaxel
Number analyzed (Participants) | 296 | 296
Percentage of participants | 11.1 [7.8 to 15.3] | 12.5 [9.0 to 16.8]
Statistical Analysis 1: Comparison: Pembrolizumab vs Paclitaxel; Stratified MN method was used for comparison of the ORR between the treatment arms. A 95% CI for the difference in response rates between the pembrolizumab arm and paclitaxel arm was provided; Test type: Other; p = 0.69010, Miettinen and Nurminen method — Stratification factors for MN method included geographic region (Europe/Israel/North America/Australia vs. Asia vs. Rest of World), TTP on first-line therapy (<6 months vs. ≥6 months), and PD-L1 status (positive vs. negative) weighting by sample size; P-value rounded to 5 decimal places; Difference in Percentage = -1.3, 95% CI 2-sided [-6.5 to 4.0]

15. Secondary Outcome: ORR According to RECIST 1.1 Based on Investigator Assessment in PD-L1 Positive Participants
Description: ORR was defined as the percentage of the participants in the analysis population who had a confirmed CR (disappearance of all non-nodal target lesions and any pathological lymph nodes must have become normal) or PR (at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD) according to RECIST 1.1 and based on investigator assessment. ORR was analyzed using the stratified Miettinen and Nurminen method, and reported with 95% CI for PD-L1 positive participants by treatment group.
Time Frame: Up to 30 months (through database cut-off date of 26 Oct 2017)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab | Paclitaxel
Number analyzed (Participants) | 196 | 199
Percentage of participants | 17.3 [12.3 to 23.4] | 15.6 [10.8 to 21.4]
Statistical Analysis 1: Comparison: Pembrolizumab vs Paclitaxel; [analysis description as in outcome 14, analysis 1]; Test type: Other; p = 0.33220, Miettinen and Nurminen method — Stratification factors for MN method included geographic region (Europe/Israel/North America/Australia vs. Asia vs. Rest of World) and TTP on first-line therapy (<6 months vs. ≥6 months), weighting by sample size; P-value rounded to 5 decimal places; Difference in Percentage = 1.6, 95% CI 2-sided [-5.8 to 9.1]

16. Secondary Outcome: ORR According to RECIST 1.1 Based on Investigator Assessment in All Participants
Description: ORR was defined as the percentage of the participants in the analysis population who had a confirmed CR (disappearance of all non-nodal target lesions and any pathological lymph nodes must have become normal) or PR (at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD) according to RECIST 1.1 and based on investigator assessment. ORR was analyzed using the stratified Miettinen and Nurminen method, and reported with 95% CI for all participants by treatment group.
Time Frame: Up to 30 months (through database cut-off date of 26 Oct 2017)
Population: All randomized participants. Participants were included in the treatment group to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab | Paclitaxel
Number analyzed (Participants) | 296 | 296
Percentage of participants | 12.2 [8.7 to 16.4] | 15.2 [11.3 to 19.8]
Statistical Analysis 1: Comparison: Pembrolizumab vs Paclitaxel; Stratified Miettinen and Nurminen's method was used for comparison of the ORR between the treatment arms. A 95% CI for the difference in response rates between the pembrolizumab arm and paclitaxel arm is provided; Test type: Other; p = 0.85922, Miettinen and Nurminen method — Stratification factors included geographic region (Europe/Israel/North America/Australia vs. Asia vs. Rest of World), TTP on first-line therapy (<6 months vs. ≥6 months), and PD-L1 status (positive vs. negative) weighting by sample size; P-value rounded to 5 decimal places; Difference in Percentage = -3.0, 95% CI 2-sided [-8.5 to 2.6]

17. Secondary Outcome: Duration of Response (DOR) According to RECIST 1.1 Based on BICR in PD-L1 Positive Participants
Description: For PD-L1 positive participants who demonstrated CR (disappearance of all non-nodal target lesions and any pathological lymph nodes must have become normal) or PR (at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD) according to RECIST 1.1 and based on BICR, DOR was defined as the time from first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first. DOR for participants who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment. DOR was analyzed using the Kaplan-Meier method and median DOR (range) in months was reported for PD-L1 positive participants with response by treatment group.
Time Frame: Up to 30 months (through database cut-off date of 26 Oct 2017)
Population: The subset of all randomized PD-L1 positive participants that showed a CR or PR according to RECIST 1.1 and based on BICR. Participants were included in the treatment group to which they were randomized.
Measure: Median (Full Range); unit: months
Arm/Group | Pembrolizumab | Paclitaxel
Number analyzed (Participants) | 31 | 27
months | 18.0 [1.4 to 26.0] | 5.2 [1.3 to 16.8]

18. Secondary Outcome: DOR According to RECIST 1.1 Based on BICR in All Participants
Description: For participants who demonstrated CR (disappearance of all non-nodal target lesions and any pathological lymph nodes must have become normal) or PR (at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD) according to RECIST 1.1 and based on BICR, DOR was defined as the time from first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first. DOR for participants who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment. DOR was analyzed using the Kaplan-Meier method and median DOR (range) in months was reported for all participants with response by treatment group.
Time Frame: Up to 30 months (through database cut-off date of 26 Oct 2017)
Population: The subset of all randomized participants that showed a CR or PR according to RECIST 1.1 and based on BICR. Participants were included in the treatment group to which they were randomized.
Measure: Median (Full Range); unit: months
Arm/Group | Pembrolizumab | Paclitaxel
Number analyzed (Participants) | 33 | 37
months | 18.0 [1.4 to 26.0] | 5.5 [1.3 to 17.7]

19. Secondary Outcome: DOR According to RECIST 1.1 Based on Investigator Assessment in PD-L1 Positive Participants
Description: For PD-L1 positive participants who demonstrated CR (disappearance of all non-nodal target lesions and any pathological lymph nodes must have become normal) or PR (at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD) according to RECIST 1.1 and based on investigator assessment, DOR was defined as the time from first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first. DOR for participants who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment. DOR was analyzed using the Kaplan-Meier method and median DOR (range) in months was reported for PD-L1 positive participants with response by treatment group.
Time Frame: Up to 30 months (through database cut-off date of 26 Oct 2017)
Population: The subset of all randomized PD-L1 positive participants that showed a CR or PR according to RECIST 1.1 and based on investigator assessment. Participants were included in the treatment group to which they were randomized.
Measure: Median (Full Range); unit: months
Arm/Group | Pembrolizumab | Paclitaxel
Number analyzed (Participants) | 34 | 31
months | 15.7 [2.7 to 23.7] | 4.3 [1.8 to 19.1]

20. Secondary Outcome: DOR According to RECIST 1.1 Based on Investigator Assessment in All Participants
Description: For participants who demonstrated CR (disappearance of all non-nodal target lesions and any pathological lymph nodes must have become normal) or PR (at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD) according to RECIST 1.1 and based on investigator assessment, DOR was defined as the time from first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first. DOR for participants who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment. DOR was analyzed using the Kaplan-Meier method and median DOR (range) in months was reported for all participants with response by treatment group.
Time Frame: Up to 30 months (through database cut-off date of 26 Oct 2017)
Population: The subset of all randomized participants that showed a CR or PR according to RECIST 1.1 and based on investigator assessment. Participants were included in the treatment group to which they were randomized.
Measure: Median (Full Range); unit: months
Arm/Group | Pembrolizumab | Paclitaxel
Number analyzed (Participants) | 36 | 45
months | 15.7 [2.7 to 23.7] | 4.3 [1.3 to 19.1]

21. Secondary Outcome: Percentage of PD-L1 Positive Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. The percentage of participants with at least one AE was reported for PD-L1 positive participants by treatment group.
Time Frame: Up to 71 months (through database cut-off date of 10 Jun 2021)
Population: All randomized PD-L1 positive participants who received at least 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Pembrolizumab | Paclitaxel
Number analyzed (Participants) | 194 | 188
Percentage of participants | 93.3 | 97.3

22. Secondary Outcome: Percentage of All Participants Who Experienced an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. The percentage of participants with at least one AE was reported for all participants by treatment group.
Time Frame: Up to 71 months (through database cut-off date of 10 Jun 2021)
Population: All randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Pembrolizumab | Paclitaxel
Number analyzed (Participants) | 294 | 276
Percentage of participants | 93.9 | 97.1
Statistical Analysis 1: Comparison: Pembrolizumab vs Paclitaxel; Between-treatment differences (Pembrolizumab vs. Paclitaxel) in the percentage of participants with events and accompanying 95% confidence intervals were based on the Miettinen and Nurminen method. Negative values correspond to a greater percentage of events for Paclitaxel; Test type: Other; Difference in Percentage = -3.2, 95% CI 2-sided [-6.9 to 0.2]

23. Secondary Outcome: Percentage of PD-L1 Positive Participants That Discontinued Study Treatment Due to AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. The percentage of participants that discontinued study treatment due to an AE was reported for PD-L1 positive participants by treatment group.
Time Frame: Up to approximately 26.4 months
Population: All randomized PD-L1 positive participants who received at least 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Pembrolizumab | Paclitaxel
Number analyzed (Participants) | 194 | 188
Percentage of participants | 4.1 | 8.0

24. Secondary Outcome: Percentage of All Participants That Discontinued Study Treatment Due to AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. The percentage of participants that discontinued study treatment due to an AE was reported for all participants by treatment group.
Time Frame: Up to approximately 26.4 months
Population: All randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Pembrolizumab | Paclitaxel
Number analyzed (Participants) | 294 | 276
Percentage of participants | 4.8 | 9.1

ADVERSE EVENTS:
Time Frame: Up to 71 months (through database cut-off date of 10 Jun 2021)
Description: All-Cause Mortality was reported for all randomized participants.
  Serious AEs and Other AEs were reported for the Safety Population: all randomized participants who received at least 1 dose of study treatment. Per protocol, disease progression of cancer on study was not considered an AE unless considered related to study drug. Therefore, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs.
Groups:
- Pembrolizumab First Course: Participants receive 200 mg IV pembrolizumab on Day 1 of each 21-day cycle, for up to 35 administrations (approximately 2 years).
- Pembrolizumab Second Course: Qualified participants who received pembrolizumab as a first course and stopped the first course of pembrolizumab due to complete response (CR) or completed the first course of pembrolizumab and had stable disease but progressed after discontinuation, initiated a second course of pembrolizumab at the investigator's discretion for up to 17 cycles (approximately 1 year additional).
Arm/Group | Pembrolizumab First Course | Paclitaxel | Pembrolizumab Second Course
All-Cause Mortality (participants affected / at risk) | 278/296 | 287/296 | 2/3
Serious Adverse Events (participants affected / at risk) | 108/294 | 68/276 | 1/3
Other Adverse Events (participants affected / at risk) | 256/294 | 260/276 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab First Course (N=294) | Paclitaxel (N=276) | Pembrolizumab Second Course (N=3)
Anaemia (Blood and lymphatic system disorders) | 11 (14) | 5 (6) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Addison's disease (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 8 (9) | 4 (4) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 4 (4) | 0 (0)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric hypomotility (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Gastric stenosis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrosplenic fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 4 (7) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatic failure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (6) | 2 (2) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 3 (3) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 5 (7) | 4 (4) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (3) | 0 (0)
Aspergillus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Biliary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Medical device site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 9 (9) | 7 (8) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Intracranial mass (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Panic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Renal injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vascular compression (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab First Course (N=294) | Paclitaxel (N=276) | Pembrolizumab Second Course (N=3)
Anaemia (Blood and lymphatic system disorders) | 44 (56) | 68 (86) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 5 (5) | 31 (62) | 0 (0)
Hypothyroidism (Endocrine disorders) | 22 (25) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 17 (17) | 12 (12) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 40 (42) | 49 (57) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 17 (21) | 16 (17) | 1 (1)
Ascites (Gastrointestinal disorders) | 19 (19) | 12 (14) | 0 (0)
Constipation (Gastrointestinal disorders) | 56 (62) | 53 (71) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 40 (42) | 72 (104) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 18 (18) | 11 (13) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 19 (20) | 17 (22) | 0 (0)
Melaena (Gastrointestinal disorders) | 6 (6) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 65 (75) | 77 (119) | 1 (1)
Oesophageal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 7 (7) | 19 (22) | 0 (0)
Vomiting (Gastrointestinal disorders) | 49 (59) | 47 (65) | 1 (1)
Asthenia (General disorders) | 30 (41) | 38 (63) | 1 (1)
Fatigue (General disorders) | 77 (95) | 89 (132) | 1 (1)
Mucosal inflammation (General disorders) | 2 (4) | 16 (19) | 0 (0)
Oedema peripheral (General disorders) | 24 (25) | 29 (37) | 0 (0)
Pyrexia (General disorders) | 32 (40) | 30 (38) | 2 (2)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 7 (9) | 17 (21) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (2)
Alanine aminotransferase increased (Investigations) | 18 (19) | 18 (26) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 24 (26) | 16 (22) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 21 (21) | 9 (12) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (5) | 36 (70) | 0 (0)
Weight decreased (Investigations) | 22 (23) | 17 (21) | 1 (1)
White blood cell count decreased (Investigations) | 3 (6) | 19 (45) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 76 (83) | 79 (99) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (8) | 2 (21) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 19 (20) | 6 (7) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 15 (17) | 10 (11) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 (29) | 24 (46) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 33 (37) | 23 (29) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 25 (31) | 0 (0)
Dizziness (Nervous system disorders) | 14 (15) | 15 (18) | 0 (0)
Headache (Nervous system disorders) | 10 (12) | 15 (20) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 8 (8) | 42 (45) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (5) | 37 (43) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 16 (16) | 24 (26) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 28 (34) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 (27) | 19 (22) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 116 (120) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 29 (29) | 18 (25) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 29 (34) | 22 (30) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/98/NCT02370498/Prot_SAP_001.pdf